CLINICAL TRIAL: NCT07297732
Title: Exploratory Study to Investigate the Tooth Whitening and Dentin Hypersensitivity Efficacy of Two Experimental Toothpastes
Brief Title: A Study to Investigate the Tooth Whitening and Dentin Hypersensitivity Effectiveness of Two Experimental Toothpastes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 300292
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Dentin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Toothpaste 1 (Experimental): Participants will be instructed to brush the entire dentition thoroughly using Test toothpaste 1 for 2-timed minutes, twice daily (morning and evening) for 8 weeks, making sure to brush all sensitive areas of the teeth.
  Interventions: Drug: Test Toothpaste 1
- Test Toothpaste 2 (Experimental): Participants will be instructed to brush the entire dentition thoroughly using Test toothpaste 2 for 2-timed minutes, twice daily (morning and evening) for 8 weeks, making sure to brush all sensitive areas of the teeth.
  Interventions: Drug: Test Toothpaste 2
- Reference Toothpaste (Active Comparator): Participants will be instructed to brush the entire dentition thoroughly using Reference toothpaste for 2-timed minutes, twice daily (morning and evening) for 8 weeks, making sure to brush all sensitive areas of the teeth.
  Interventions: Drug: Reference Toothpaste

INTERVENTIONS:
Drug: Test Toothpaste 1 — Toothpaste containing Potassium nitrate
  Arms: Test Toothpaste 1
Drug: Test Toothpaste 2 — Toothpaste containing Potassium nitrate
  Arms: Test Toothpaste 2
Drug: Reference Toothpaste — Regular fluoride toothpaste
  Arms: Reference Toothpaste

SUMMARY:
The aim of this exploratory clinical study is to investigate the tooth whitening potential, Dentin Hypersensitivity (DH) efficacy, and oral tolerability of two experimental toothpastes in a DH population with appropriate tooth shade and dental stain levels for the evaluation of whitening performance.

DETAILED DESCRIPTION:
This will be a single center, randomized, controlled, examiner-blind, 3-treatment arm, stratified (Baseline mean VITA Bleached Guide 3D-MASTER score), parallel design, clinical study in healthy participants, aged 18-65 years inclusive, with sufficient tooth discoloration/surface stain to evaluate the whitening potential of the experimental formulations, and self-reported/clinically diagnosed dentin hypersensitivity. Participants who meet the required study criteria at Screening and Baseline will be randomized to one of three study toothpastes. Approximately 105 qualifying participants will be stratified and randomized to study treatment (approximately 35 participants per treatment group).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent before any study procedures are performed.
* Participant is biologically male or female.
* Participant is 18 to 65 years of age, inclusive, at the time of signing the consent form.
* Participant is willing and able to comply with the study visit schedule, product usage instructions, lifestyle restrictions and other study procedures.
* Participant is in good general, oral and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in self-reported medical history (example, a medical condition confirmed to be causing xerostomia), or upon oral examination, that would impact their safety or wellbeing, or the outcomes of the study, if they were to participate in the study, or affect their ability to understand and follow study requirements.
* Participant must have History of tooth sensitivity lasting more than six months but not more than 10 years (self-reported) and must have good general oral health, with a minimum of 20 natural teeth.
* Participant must have minimum of 2 accessible, non-adjacent teeth (incisors, canines, premolars), in different quadrants

Exclusion Criteria:

* Participant is an employee of the study site directly involved in the conduct of the study, or an employee of the study site otherwise supervised by the investigator, or a member of their immediate family.
* Participant is an employee of the sponsor directly involved in the conduct of the study or a member of their immediate family.
* Female participant who is pregnant (self-reported) or intending to become pregnant during the study (self-reported) or who is who is breastfeeding (self-reported).
* Participant with known or suspected intolerance or hypersensitivity to any of the study products (Acclimatization Toothpaste or study toothpastes), any of their stated ingredients or closely related compounds (self-reported).
* Participant with a recent history (within the last year) of alcohol or other substance abuse (self-reported).
* Participant is participating in, or has participated in, other studies (including non-medicinal studies) involving an investigational product (IP) within 30 days of Screening (Visit 1) or plans to participate in other studies (including non-medicinal studies) during this study (self-reported).
* Participant has participated in a tooth sensitivity study within 8 weeks of Screening (Visit 1) (self-reported).
* Participant is currently using an oral care product indicated for DH relief or care of sensitive teeth or has used an anti-hypersensitivity oral care product within 8 weeks of Screening (Visit 1) (self-reported).
* Participant is currently using an oral care product primarily intended for tooth whitening benefits or has used such a product within 8 weeks of Screening (Visit 1) (self-reported).
* Participant has had professional tooth de-sensitizing treatment within 8 weeks of Screening (Visit 1) (self-reported).
* Participant is taking daily doses of medications/treatments (self-reported) which, in the opinion of the investigator or medically qualified designee, could interfere with their perception of tooth sensitivity (example, analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilizers, antidepressants, mood-altering and anti-inflammatory drugs).
* Participant is taking daily doses of a medication (self-reported) which, in the opinion of the investigator or medically qualified designee, is causing xerostomia.
* Participant requires antibiotic prophylaxis for dental procedures (self-reported).
* Participant has had a tooth whitening procedure (professional or in-home treatment) within 12 months of Screening (Visit 1) (self-reported).
* Participant has had dental prophylaxis within 8 weeks of Screening (Visit 1) (self-reported).
* Participant has had treatment for periodontal disease (including surgery) within 12 months of Screening (Visit 1) (self-reported).
* Participant has had scaling or root planing within 3 months of Screening (Visit 1) (self-reported).
* Participant with, in the opinion of the investigator or medically qualified designee, gross periodontal disease.
* Participant with a tongue or lip piercing.
* Participant with, in the opinion of the investigator or medically qualified designee, evidence of gross intra-oral neglect or the need for extensive dental therapy.
* Participant with evidence of current/recent active dental caries or (self-reported) treatment for decay within 12 months of Screening (Visit 1).
* Participant with a fixed or removable partial prosthesis, multiple dental implants, fixed or removable orthodontic braces/bands and/or a fixed orthodontic retainer which, in the opinion of the investigator or dentally qualified designee, could impact study outcomes.
* Specific dentition exclusions: For eligible teeth (DH assessment)

  1. Tooth with evidence of current/recent caries.
  2. Tooth with treatment for decay within 12 months of Screening (Visit 1) (self-reported).
  3. Tooth with exposed dentin and deep, defective or facial restorations.
  4. Tooth with a full crown or veneer.
  5. Tooth adjacent to a bridge abutment or crown which, in the opinion of the investigator or dentally qualified designee, could impact study outcomes.
  6. Sensitive tooth with contributing etiologies other than EAR to exposed dentin.
  7. Sensitive tooth not expected to benefit from use of an anti-hypersensitivity toothpaste, in the opinion of the investigator or dentally qualified designee.
* Participant has taken antibiotics in the 2 weeks prior to Screening (Visit 1) (self-reported).
* Participant has taken antibiotics in the 2 weeks prior to Baseline (Visit 2), that is, during the 2-week Acclimatization Period (self-reported).
* Participant has previously been enrolled in this study.
* Participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Mean VITA Shade Score at Baseline, Weeks 1, 2, 4 and 8 | Baseline, Weeks 1, 2, 4 and 8
  Tooth color of the facial surfaces of the six anterior maxillary teeth will be visually assessed using the VITA Bleachedguide 3D-MASTER shade guide. It consists of a value-ranked ordered scale from 1 (lightest) to 29 (darkest). The shade of each assessable tooth surface/region will be scored by the clinical examiner with reference to the guide, where lower score indicates improvement.
Mean Total Modified Lobene Stain Index (MLSI) Score at Baseline, Weeks 1, 2, 4 and 8 | Baseline, Weeks 1, 2, 4 and 8
  Dental stain will be visually assessed for the facial surfaces of the teeth (incisors and canines) using the MLSI. For each tooth surface assessed, Area (A) and Intensity (I) of dental stain will be scored separately on the scale of 0 to 3 and the mean total score will be presented, where 0=Area with no stain, 1=Stain covering up to one third of area and light intensity stain, 2=Stain covering up to two thirds of area and moderate intensity stain, 3=Stain covering more than two thirds of area and heavy intensity stain. Total MLSI score = Area score multiplied by Intensity score and ranging from 0 to 9, where lower score indicates improvement.

SECONDARY OUTCOMES:
Schiff Sensitivity Score at Baseline, Week 4 and Week 8 | Baseline, Week 4 and 8
  Evaporative (air) sensitivity will be assessed by participant's response to an evaporative (air) stimulus after stimulation of 2 selected test teeth. Response of participant will be scored using Schiff sensitivity scale which ranges from 0-3, where 0=Does not respond to air stimulation; 1=Responds to air stimulus but does not request discontinuation of stimulus; 2=Responds to air stimulus and requests discontinuation or moves from stimulus; 3=Responds to stimulus, considers stimulus to be painful and requests discontinuation of the stimulus. The lower score indicates improvement.
Tactile Threshold at Baseline, Week 4 and Week 8 | Baseline, Week 4 and 8
  The tactile sensitivity will be assessed by administrating a constant pressure using a Yeaple probe. The tactile threshold is the maximum pressure applied without the participant reporting pain or discomfort. The tactile threshold for 2 selected test teeth will be determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gives two consecutives 'yes' responses will be recorded as the tactile threshold. The greater the tactile threshold, the less sensitive the tooth.

CONTACTS AND LOCATIONS:
Locations (1):
- Silverstone Research Group, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.